CLINICAL TRIAL: NCT02145468
Title: A Clinical Outcomes Study to Compare the Incidence of Major Adverse Cardiovascular Events in Subjects Presenting With Acute Coronary Syndrome Treated With Losmapimod Compared to Placebo (PM1116197) LosmApimod To Inhibit p38 MAP Kinase as a TherapeUtic Target and moDify Outcomes After an Acute Coronary syndromE (LATITUDE)-TIMI 60.
Brief Title: A Phase 3 Clinical Outcomes Study to Compare the Incidence of Major Adverse Cardiovascular Events in Subjects Presenting With Acute Coronary Syndrome Treated With Losmapimod Compared to Placebo (LATITUDE-TIMI 60)
Acronym: LATITUDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: The TIMI Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116197
Record Dates: First submitted 2014-05-15; First posted 2014-05-23 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-03

CONDITIONS: Acute Coronary Syndrome
Keywords: Myocardial infarction; Acute coronary syndrome; Cardiovascular disease; p38 mitogen-activated protein kinase (MAPK) inhibitor; NSTEMI; Losmapimod; STEMI
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Cardiovascular Diseases; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Losmapimod (Experimental): Losmapimod 7.5 mg twice daily oral tablet
  Interventions: Drug: Losmapimod 7.5 mg twice daily; Drug: Standard therapy
- Placebo (Placebo Comparator): Placebo twice daily oral tablet
  Interventions: Drug: Placebo twice daily; Drug: Standard therapy

INTERVENTIONS:
Drug: Losmapimod 7.5 mg twice daily — Subjects will receive Losmapimod 7.5 mg as film-coated, round, plain faced tablets.
  Other Names: GW856553
  Arms: Losmapimod
Drug: Placebo twice daily — Subjects will receive placebo as film-coated, round, plain faced tablets.
  Arms: Placebo
Drug: Standard therapy — Subjects will receive standard therapy consistent with the appropriate guidelines from professional societies. The standard therapy includes nitrates, morphine sulfate, beta adrenergic blockers, renin-angiotensin aldosterone inhibitors, other anti-ischemic therapies, and analgesic therapy.

SUMMARY:
Losmapimod is a new anti-inflammatory medication which potentially may benefit patients with Acute Coronary Syndrome, (ACS), a condition which includes heart attack. There is a growing understanding that the inflammatory response to ACS is integral to the subsequent evolution of plaque instability. Losmapimod inhibits p38 mitogen activated protein kinase (MAPK), an enzyme which may play a central role in inflammation in the setting of heart attack. Inhibition of p38 MAPK may stabilize atherosclerotic plaques, reduce the risk of subsequent plaque rupture, indirectly improve vascular function and prevent subsequent thrombosis, and thus reduce infarct size and the risk of subsequent cardiac events. This study will test whether losmapimod can safely reduce the risk of a subsequent cardiovascular event (such as death, heart attack, or near heart attack requiring urgent treatment ) when started immediately after ACS (specifically, heart attack). Patients who present with heart attack and qualify for the study will be randomly assigned to receive 3 months treatment with either losmapimod twice daily or placebo, which will be administered in addition to the usual standard of care therapies for heart attack. Following the in-hospital period, subjects will return for outpatient visits at 4 and 12 weeks, as well as a follow up visit at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Men or women at least 35 years old. Women must be post-menopausal or using a highly effective method for avoidance of pregnancy
* Hospitalization for NSTEMI or STEMI (Universal Definition Type 1 MI)
* With the following timing of symptoms: NSTEMI: Presence of ischemic symptoms (>=5 minutes) at rest within 24 hours prior to randomization (may include qualifying episode). STEMI: Onset of qualifying ischemic symptoms within 12 hours of randomization.
* At least one of the following
* Age >=60 years at randomization.
* Myocardial infarction prior to the qualifying ACS event
* CABG prior to qualifying ACS event.
* NSTEMI with new ischemic ST-segment depression >= 0.1 mV in >= 2 contiguous leads.
* Diabetes mellitus requiring pharmacotherapy.
* Coexistent clinically diagnosed arterial disease

Exclusion Criteria:

* Unable to be randomized prior to coronary revascularization or fibrinolysis for the qualifying MI.
* Current severe heart failure or shock
* Ongoing clinical instability
* History of chronic liver disease
* Known severe renal impairment
* Any condition, other than vascular disease, with life expectancy <1 year that might prevent the subject from completing the study.
* Known active tuberculosis, HIV, active opportunistic or life threatening infections.
* Vaccination with a live attenuated vaccine within 6 weeks of randomization.
* Concomitant use of cytotoxic chemotherapy for cancer or known ongoing or anticipated use of chronic severe immunosuppressive agents
* Positive pregnancy test or is known to be pregnant or lactating
* Known alcohol or drug abuse within the past 6 months
* Any current mental condition, which may affect study compliance or prevent understanding of the aims, investigational procedures or possible consequences of the study.
* Participation in a study of an investigational medication within the past 30 days.
* Anticipated inability to comply with any study procedures, including participation in study visits according to the visit schedule through 24 weeks.
* Use of another investigational product within 30 days or 5 half-lives (whichever is longer) or according to local regulations, or currently participating in a study of an investigational device. Subjects must be randomized only one time in this investigational study
* Any other reason the investigator deems the subject to be unsuitable for the study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3503 (Actual)
Dates: Start 2014-06-03 (Actual); Primary Completion 2015-12-14 (Actual); Study Completion 2015-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (305):
- United States (86):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Cottonwood, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Monterey, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Jacksonville Beach, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Rome, Georgia
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Aurora, Illinois
  - GSK Investigational Site, Elmhurst, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Muncie, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, Alexandria, Louisiana
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Zachary, Louisiana
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Grand Blanc, Michigan
  - GSK Investigational Site, Marquette, Michigan
  - GSK Investigational Site, Rochester, Michigan
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Duluth, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Flemington, New Jersey
  - GSK Investigational Site, Ridgewood, New Jersey
  - GSK Investigational Site, Teaneck, New Jersey
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Poughkeepsie, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Mansfield, Ohio
  - GSK Investigational Site, Zanesville, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Abington, Pennsylvania
  - GSK Investigational Site, Chambersburg, Pennsylvania
  - GSK Investigational Site, Danville, Pennsylvania
  - GSK Investigational Site, Doylestown, Pennsylvania
  - GSK Investigational Site, Wilkes-Barre, Pennsylvania
  - GSK Investigational Site, York, Pennsylvania
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Round Rock, Texas
  - GSK Investigational Site, Victoria, Texas
  - GSK Investigational Site, Roanoke, Virginia
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Morgantown, West Virginia
  - GSK Investigational Site, Manitowoc, Wisconsin
  - GSK Investigational Site, Wausau, Wisconsin
- Argentina (6):
  - GSK Investigational Site, Quilmes, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Venado Tuerto, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Corrientes
  - GSK Investigational Site, Santa Fe
- Australia (10):
  - GSK Investigational Site, Brisbane, Queensland
  - GSK Investigational Site, Cairns, Queensland
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Nambour, Queensland
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Epping, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Murdoch, Western Australia
  - GSK Investigational Site, Nedlands, Western Australia
- Belgium (10):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Brasschaat
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Mechelen
  - GSK Investigational Site, Yvoir
- Bulgaria (4):
  - GSK Investigational Site, Blagoevgrad
  - GSK Investigational Site, Dimitrovgrad
  - GSK Investigational Site, Pazardzhik
  - GSK Investigational Site, Sofia
- Canada (9):
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Scarborough Village, Ontario
  - GSK Investigational Site, Thunder Bay, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Chile (4):
  - GSK Investigational Site, Temuco, Región de La Araucania
  - GSK Investigational Site, Concepción, Región Del Biobio
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Czechia (9):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, České Budějovice
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Liberec
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Ústí nad Labem
  - GSK Investigational Site, Zlín
- Denmark (4):
  - GSK Investigational Site, Hellerup
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, København NV
  - GSK Investigational Site, København S
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (10):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Montauban
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pau
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tourcoing
  - GSK Investigational Site, Valenciennes
- Germany (21):
  - GSK Investigational Site, Bad Krozingen, Baden-Wurttemberg
  - GSK Investigational Site, Esslingen am Neckar, Baden-Wurttemberg
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Bernau bei Berlin, Brandenburg
  - GSK Investigational Site, Bad Nauheim, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Giessen, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Langen, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Leverkusen, North Rhine-Westphalia
  - GSK Investigational Site, Mönchengladbach, North Rhine-Westphalia
  - GSK Investigational Site, Wuppertal, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Hamburg
- Greece (5):
  - GSK Investigational Site, Alexandroupoli
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Chalcis
  - GSK Investigational Site, N. Efkarpia, Thessaloniki
  - GSK Investigational Site, Thessaloniki
- Hong Kong (3):
  - GSK Investigational Site, Chai Wan
  - GSK Investigational Site, Kowloon
  - GSK Investigational Site, Shatin, New Territories
- Hungary (4):
  - GSK Investigational Site, Balatonfüred
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Szolnok
  - GSK Investigational Site, Zalaegerszeg
- Israel (5):
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Haddera
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Nahariya
  - GSK Investigational Site, Tel Aviv
- Italy (6):
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Cremona, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Perugia, Umbria
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Querétaro
  - GSK Investigational Site, San Luis Potosí City
- Netherlands (14):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Delft
  - GSK Investigational Site, Deventer
  - GSK Investigational Site, Helmond
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Schiedam
  - GSK Investigational Site, Sittard-geleen
  - GSK Investigational Site, Tilburg
  - GSK Investigational Site, Venlo
  - GSK Investigational Site, Zwolle
- New Zealand (6):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Grafton, Auckland
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, New Plymouth
  - GSK Investigational Site, Otahuhu, Auckland
  - GSK Investigational Site, Wellington South
- Norway (5):
  - GSK Investigational Site, Lillehammer
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Skien
  - GSK Investigational Site, Stavanger
  - GSK Investigational Site, Tromsø
- Philippines (4):
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Pasig
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, San Juan City
- Poland (12):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Inowrocław
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lubin
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wałbrzych
  - GSK Investigational Site, Wroclaw
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Craiova
- Russia (13):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Gatchina
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Tyumen
- Slovakia (4):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Martin
  - GSK Investigational Site, Nitra
- South Africa (6):
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Kuils River
  - GSK Investigational Site, Parktown West
  - GSK Investigational Site, Pinelands
  - GSK Investigational Site, Somerset West
- South Korea (4):
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Ganwon-do
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Seoul
- Spain (8):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Galdakano
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
- Sweden (7):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Helsingborg
  - GSK Investigational Site, Jönköping
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Östersund
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Västerås
- Taiwan (4):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Hualien City
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taipei
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- Ukraine (7):
  - GSK Investigational Site, Cherkassy
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Uzhhorod
  - GSK Investigational Site, Zaporizhzhya
- United Kingdom (6):
  - GSK Investigational Site, Basingstoke
  - GSK Investigational Site, Bournemouth
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, York

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Cavender MA, O'Donoghue ML, Abbate A, Aylward P, Fox KA, Glaser RX, Park JG, Lopez-Sendon J, Steg PG, Sabatine MS, Morrow DA. Inhibition of p38 MAP kinase in patients with ST-elevation myocardial infarction - findings from the LATITUDE-TIMI 60 trial. Am Heart J. 2022 Jan;243:147-157. doi: 10.1016/j.ahj.2021.08.022. Epub 2021 Sep 8. PMID 34508693
- [Derived] O'Donoghue ML, Glaser R, Cavender MA, Aylward PE, Bonaca MP, Budaj A, Davies RY, Dellborg M, Fox KA, Gutierrez JA, Hamm C, Kiss RG, Kovar F, Kuder JF, Im KA, Lepore JJ, Lopez-Sendon JL, Ophuis TO, Parkhomenko A, Shannon JB, Spinar J, Tanguay JF, Ruda M, Steg PG, Theroux P, Wiviott SD, Laws I, Sabatine MS, Morrow DA; LATITUDE-TIMI 60 Investigators. Effect of Losmapimod on Cardiovascular Outcomes in Patients Hospitalized With Acute Myocardial Infarction: A Randomized Clinical Trial. JAMA. 2016 Apr 19;315(15):1591-9. doi: 10.1001/jama.2016.3609. PMID 27043082
- [Derived] O'Donoghue ML, Glaser R, Aylward PE, Cavender MA, Crisp A, Fox KA, Laws I, Lopez-Sendon JL, Steg PG, Theroux P, Sabatine MS, Morrow DA. Rationale and design of the LosmApimod To Inhibit p38 MAP kinase as a TherapeUtic target and moDify outcomes after an acute coronary syndromE trial. Am Heart J. 2015 May;169(5):622-630.e6. doi: 10.1016/j.ahj.2015.02.012. Epub 2015 Feb 23. PMID 25965709
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 116197 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116197 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116197 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116197 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116197 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116197 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116197 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned in 2 parts (Part A, N=3500 and Part B, N=22000). Upon completing Part A, a decision was made not to progress to Part B because of lack of efficacy. 3503 participants were randomized to Part A, 14 participants were excluded due to concerns over data integrity. 3489 participants were analyzed.
Pre-assignment Details: Eligible: >=35 years and hospitalized with type1 myocardial infarction (MI) and 1 additional predictor of cardiovascular (CV) risk; Excluded: unstable, known liver disease, life-threatening/opportunistic infection, severe renal impairment, NYHA III/IV or Killip III/IV CHF. All participants were followed until they withdrew consent to participate.
Groups:
- Placebo: Participants received losmapimod matching placebo tablets via oral route, twice daily (BID), according to the randomization schedule for 12 weeks in addition to standard of care, and were followed for an additional 12 weeks after completing treatment, for a total study duration of 24 weeks.
- Losmapimod 7.5 Mllligrms BID: Participants received losmapimod 7.5 milligrams (mg) tablets via oral route, BID, according to the randomization schedule for 12 weeks in addition to standard of care, and were followed for an additional 12 weeks after completing treatment, for a total study duration of 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Losmapimod 7.5 Mllligrms BID
Started | 1758 | 1731
Completed | 1753 | 1723
Not Completed | 5 | 8
Not completed — Withdrawal by Subject | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received losmapimod matching placebo tablets via oral route, BID, according to the randomization schedule for 12 weeks in addition to standard of care, and were followed for an additional 12 weeks after completing treatment, for a total study duration of 24 weeks.
- Losmapimod 7.5 mg BID: Participants received losmapimod 7.5 mg tablets via oral route, BID, according to the randomization schedule for 12 weeks in addition to standard of care, and were followed for an additional 12 weeks after completing treatment, for a total study duration of 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Losmapimod 7.5 mg BID | Total
Number analyzed (Participants) | 1758 | 1731 | 3489
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (9.72) | 66.7 (10.00) | 66.6 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 532 | 500 | 1032
  Male | 1226 | 1231 | 2457
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 8 | 16
  Asian | 99 | 105 | 204
  Native Hawaiian or Other Pacific Islander | 5 | 10 | 15
  Black or African American | 25 | 20 | 45
  White | 1616 | 1585 | 3201
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of Major Adverse Cardiovascular Events (MACE) Through Week 12
Description: The primary efficacy endpoint is the composite measure of adjudicated MACE that includes the time to first occurrence of CV death (death due to a cardiovascular cause), MI or SRI-UR (Severe Recurrent Ischemia requiring Urgent coronary artery Revascularization). Death for which the Clinical Events Committee (CEC) or investigator were unable to establish cause were analyzed as CV deaths.
Time Frame: Up to 12 weeks
Population: Intent-To-Treat (ITT) Population. ITT population comprised of all randomized participants.
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  First occurence of MACE | 123 | 139
  CV Death | 34 | 31
  MI | 74 | 90
  SRI-UR | 15 | 18
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Test type: Superiority; p = 0.238, Log Rank; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.91 to 1.47] — Hazard ratio and CI are estimated using a Cox proportional hazard regression model stratified by baseline STEMI/NSTEMI status with treatment as the only covariate. A hazard ratio <1 indicates a lower risk with the treatment compared with placebo

2. Secondary Outcome: Number of Participants With First Occurrence of MACE Through Week 24
Description: Number of participants with first occurrence of MACE through Week 24 including CV death, MI or SRI-UR are presented. Death for which the CEC or investigator were unable to establish cause were analyzed as CV deaths.
Time Frame: Up to Week 24
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  First occurrence of MACE | 162 | 176
  CV Death | 45 | 38
  MI | 98 | 117
  SRI-UR | 19 | 21
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Test type: Superiority; p = 0.329, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.90 to 1.38] — Hazard ratio and CI are estimated using a Cox proportional hazard regression model stratified by baseline STEMI/NSTEMI status with treatment as the only covariate. A hazard ratio <1 indicates a lower risk. with the treatment compared with placebo

3. Secondary Outcome: Number of Participants With First Occurrence of the Composite of CV Death or MI up to Week 12 and Week 24
Description: Week 12 results are considered the principal secondary endpoint. Number of participants with first occurrence of the composite of CV death or MI up to Week 12 and Week 24 are summarized.
Time Frame: Week 12 and Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 110 | 122
  Week 24 | 145 | 156
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; CV death or MI, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.338, Log Rank; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.88 to 1.47] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 7.5 mg BID; CV death or MI, Placebo Vs Losmapimod 7.5 mg BID at Week 24; Test type: Superiority; p = 0.410, Log Rank; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.88 to 1.38] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With First Occurrence of the Composite of CV Death, MI or Hospitalization for Heart Failure (HF) up to Week 12 and Week 24.
Description: Number of participants with first occurrence of the composite of CV death, MI or hospitalization for HF up to Week 12 and Week 24 are presented.
Time Frame: Week 12 and Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 131 | 140
  Week 24 | 169 | 178
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; CV death, MI or hospitalization for HF, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.472, Log Rank; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.86 to 1.38] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With First Occurrence of the Expanded Composite of Arterial CV Events Defined as CV Death, MI, SRI-UR or Stroke Through to Week 12 and Week 24
Description: Number of participants with first occurrence of the expanded composite of arterial CV events defined as CV death, MI, SRI-UR or stroke through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 135 | 151
  Week 24 | 174 | 190
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Composite of arterial CV events (CV death, MI, SRI-UR or stroke), Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.91 to 1.44] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants With First Occurrence of the Composite of Coronary Events Defined as CHD Death, MI, SRI-UR or Any Unplanned Coronary Artery Revascularization Through to Week 12 and Week 24
Description: Number of participants with first occurrence of the composite of coronary events defined as coronary heart disease (CHD) death, MI, SRI-UR or any unplanned coronary artery revascularization through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 144 | 152
  Week 24 | 186 | 194
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Composite of coronary events (CHD death, MI, SRI-UR or any unplanned coronary artery revascularization), Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.505, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.86 to 1.36] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants With First Occurrence of the Composite of CV Death or Hospitalization for HF Through to Week 12 and Week 24
Description: Number of participants with first occurrence of the composite of CV death or hospitalization for HF through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 72 | 64
  Week 24 | 94 | 86
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Composite of CV death or hospitalization for HF, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.536, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.64 to 1.26] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 7.5 mg BID; Composite of CV death or hospitalization for HF, Placebo Vs Losmapimod 7.5 mg BID at Week 24; Test type: Superiority; p = 0.6, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.69 to 1.24] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Number of Participants With First Occurrence of the Composite of CV Death, MI or Stroke Through to Week 12 and Week 24
Description: Number of participants with first occurrence of the composite of CV death, MI or stroke through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 122 | 134
  Week 24 | 157 | 170
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Composite of CV death, MI or stroke, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.356, Log Rank; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.88 to 1.43] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Number of Participants With First Occurrence of the Expanded Composite of CV Death, MI, SRI-UR, Stroke or Hospitalization for HF Through to Week 12 and Week 24
Description: Number of participants with first occurrence of the expanded composite of CV death, MI, SRI-UR, stroke or hospitalization for HF through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 155 | 169
  Week 24 | 197 | 212
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Composite of CV death, MI, SRI-UR, stroke or hospitalization for HF, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.329, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.9 to 1.39] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Number of Participants With First Occurrence of the Composite of CHD Death, MI or SRI-UR Through to Week 12 and Week 24
Description: Number of participants with first occurrence of the composite of CHD death, MI or SRI-UR through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 119 | 133
  Week 24 | 152 | 167
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Composite of CHD death, MI or SRI-UR, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.285, Log Rank; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.89 to 1.47] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Number of Participants With First Occurrence of the Composite of CHD Death or MI Through to Week 12 and Week 24
Description: Number of participants with first occurrence of the composite of CHD death or MI through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 106 | 116
  Week 24 | 135 | 147
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Composite of CHD death or MI, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.401, Log Rank; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.86 to 1.46] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Number of Participants With First Occurrence of the Composite of All-cause Death, MI or SRI-UR Through to Week 12 and Week 24
Description: Number of participants with first occurrence of the composite of all-cause death, MI or SRI-UR through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 128 | 142
  Week 24 | 169 | 185
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Composite of all-cause death, MI or SRI-UR,Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.295, Log Rank; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.89 to 1.44] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Number of Participants With First Occurrence of the Composite of All-cause Death or MI Through to Week 12 and Week 24
Description: Number of participants with first occurrence of the composite of all-cause death or MI through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 115 | 125
  Week 24 | 152 | 165
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Composite of all-cause death or MI, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.412, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.86 to 1.43] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Number of Participants With First Occurrence of the Composite of CV Death, Type I (Spontaneous) MI or SRI-UR Through to Week 12 and Week 24
Description: Number of participants with first occurrence of the composite of CV death, type I (spontaneous) MI or SRI-UR through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 86 | 94
  Week 24 | 122 | 127
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Composite of CV death, type I (spontaneous) MI or SRI-UR, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.469, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.83 to 1.49] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Number of Participants With First Occurrence of the Composite of CV Death or Type I (Spontaneous) MI Through to Week 12 and Week 24
Description: Number of participants with first occurrence of the composite of CV death or type I (spontaneous) MI through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 73 | 77
  Week 24 | 104 | 106
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Composite of CV death or type I (spontaneous) MI, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.664, Log Rank; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.78 to 1.48] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Number of Participants With First Occurrence of Definite or Probable Stent Thrombosis Through to Week 12 and Week 24
Description: Number of participants with first occurrence of definite or probable stent thrombosis through to Week 12 and Week 24 are presented. Participants receiving stent prior to randomization or during the study prior to Week 12 were included.
Time Frame: Week 12, Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, in the category titles).
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12, n=1281, 1306 | 19 | 11
  Week 24, n=1758, 1731 | 21 | 12
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Participants with first occurrence of definite or probable stent thrombosis, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.130, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.27 to 1.19] — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: Number of Participants Re-hospitalized Within 30 Days of Discharge
Description: Participants who had a death or re-hospitalization within 30 days of discharge, plus participants who were never discharged from the initial hospitalization were included.
Time Frame: Within up to 30 days of post discharge
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants | 210 | 213
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Test type: Superiority; p = 0.744, Wald chi-squared; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.84 to 1.27] — Odds ratio is estimated using a logistic regression model stratified by baseline STEMI/NSTEMI status with treatment as the only covariate. An odds ratio <1 indicates a lower risk with the treatment compared with placebo

18. Secondary Outcome: Number of Participants With All-cause Mortality Through to Week 12 and Week 24
Description: Number of participants with all-cause mortality through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 49 | 39
  Week 24 | 68 | 57
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Participants with all-cause mortality, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.309, Log Rank; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.53 to 1.22] — [estimate comment as in outcome 1, analysis 1]

19. Secondary Outcome: Number of Participants With CV Death Events Through to Week 12 and Week 24
Description: Number of participants with CV death events through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 44 | 36
  Week 24 | 59 | 47
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; CV death events, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.398, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.53 to 1.28] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 7.5 mg BID; CV death events, Placebo Vs Losmapimod 7.5 mg BID at Week 24; Test type: Superiority; p = 0.264, Log Rank; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.55 to 1.18] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Number of Participants With CHD Death Events Through to Week 12 and Week 24
Description: Number of participants with CHD death events through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 40 | 30
  Week 24 | 49 | 37
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; CHD death events, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.251, Log Rank; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.47 to 1.22] — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: Number of Participants With First Occurrence of Myocardial Infarction (Fatal and Non-fatal) Events Through to Week 12 and Week 24
Description: Number of participants with first occurrence of myocardial infarction (fatal and non-fatal) events through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 75 | 90
  Week 24 | 99 | 117
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Myocardial infarction (fatal and non-fatal) events, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.182, Log Rank; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.91 to 1.67] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 7.5 mg BID; Myocardial infarction (fatal and non-fatal) events, Placebo Vs Losmapimod 7.5 mg BID at Week 24; Test type: Superiority; p = 0.158, Log Rank; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.93 to 1.58] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Number of Participants With First Occurrence of Type I (Spontaneous) MI Events Through to Week 12 and Week 24
Description: Number of participants with first occurrence of type I (spontaneous) MI events through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 32 | 42
  Week 24 | 51 | 62
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Type I (spontaneous) MI events, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.21, Log Rank; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.85 to 2.12] — [estimate comment as in outcome 1, analysis 1]

23. Secondary Outcome: Number of Participants With First Occurrence of SRI-UR Events Through to Week 12 and Week 24
Description: Number of participants with first occurrence of SRI-UR events through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 16 | 18
  Week 24 | 22 | 22
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; SRI-UR events, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.697, Log Rank; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.58 to 2.24] — [estimate comment as in outcome 1, analysis 1]

24. Secondary Outcome: Number of Participants With First Occurrence of Stroke (Fatal and Non-fatal) Events Through to Week 12 and Week 24
Description: Number of participants with first occurrence of stroke (fatal and non-fatal) events through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 15 | 14
  Week 24 | 19 | 18
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Stroke (fatal and non-fatal) events, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.883, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.46 to 1.96] — [estimate comment as in outcome 1, analysis 1]

25. Secondary Outcome: Number of Participants With First Occurrence of Hospitalization for HF Through to Week 12 and Week 24
Description: Number of participants with first occurrence of hospitalization for HF through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 42 | 35
  Week 24 | 53 | 49
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Hospitalization for HF, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.457, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.54 to 1.32] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Losmapimod 7.5 mg BID; Hospitalization for HF, Placebo Vs Losmapimod 7.5 mg BID at Week 24; Test type: Superiority; p = 0.736, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.63 to 1.38] — [estimate comment as in outcome 1, analysis 1]

26. Secondary Outcome: Number of Participants With First Occurrence of Any Unplanned Coronary Revascularization Through to Week 12 and Week 24
Description: Number of participants with first occurrence of any unplanned coronary revascularization through to Week 12 and Week 24 are presented.
Time Frame: Week 12, Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Losmapimod 7.5 mg BID
Number analyzed (Participants) | 1758 | 1731
Participants
  Week 12 | 57 | 62
  Week 24 | 75 | 87
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 7.5 mg BID; Any unplanned coronary revascularization, Placebo Vs Losmapimod 7.5 mg BID at Week 12; Test type: Superiority; p = 0.581, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.77 to 1.59] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until follow-up (up to Week 24)
Description: SAEs and AEs are reported for the Safety population which comprised of all randomized participants who had received at least one dose of investigational product (IP). The SAEs are all SAEs excluding positively CEC-adjudicated CV events.
Arm/Group | Placebo | Losmapimod 7.5 mg BID
All-Cause Mortality (participants affected / at risk) | 68/1752 | 57/1724
Serious Adverse Events (participants affected / at risk) | 323/1752 | 363/1724
Other Adverse Events (participants affected / at risk) | 370/1752 | 376/1724
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1752) | Losmapimod 7.5 mg BID (N=1724)
Angina unstable (Cardiac disorders) | 24 | 26
Angina pectoris (Cardiac disorders) | 14 | 24
Atrial fibrillation (Cardiac disorders) | 14 | 19
Acute myocardial infarction (Cardiac disorders) | 7 | 13
Cardiac failure (Cardiac disorders) | 6 | 10
Cardiac failure congestive (Cardiac disorders) | 5 | 8
Ventricular fibrillation (Cardiac disorders) | 5 | 7
Ventricular tachycardia (Cardiac disorders) | 5 | 7
Cardiogenic shock (Cardiac disorders) | 6 | 5
Atrial flutter (Cardiac disorders) | 4 | 4
Cardiac arrest (Cardiac disorders) | 3 | 5
Atrioventricular block complete (Cardiac disorders) | 4 | 3
Sinus node dysfunction (Cardiac disorders) | 4 | 3
Pericardial effusion (Cardiac disorders) | 2 | 3
Coronary artery perforation (Cardiac disorders) | 2 | 2
Pericarditis (Cardiac disorders) | 3 | 1
Arteriospasm coronary (Cardiac disorders) | 1 | 2
Bradycardia (Cardiac disorders) | 0 | 3
Cardiac tamponade (Cardiac disorders) | 1 | 2
Coronary artery disease (Cardiac disorders) | 0 | 3
Coronary artery dissection (Cardiac disorders) | 3 | 0
Myocardial ischaemia (Cardiac disorders) | 3 | 0
Palpitations (Cardiac disorders) | 1 | 1
Torsade de pointes (Cardiac disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Aortic valve disease (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Coronary artery thrombosis (Cardiac disorders) | 1 | 0
Dressler's syndrome (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial rupture (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Pericarditis lupus (Cardiac disorders) | 1 | 0
Postinfarction angina (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular dyssynchrony (Cardiac disorders) | 0 | 1
Ventricular flutter (Cardiac disorders) | 1 | 0
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 12 | 16
Sepsis (Infections and infestations) | 4 | 4
Urinary tract infection (Infections and infestations) | 3 | 5
Cystitis (Infections and infestations) | 2 | 3
Gastroenteritis (Infections and infestations) | 1 | 4
Urosepsis (Infections and infestations) | 2 | 3
Bronchitis (Infections and infestations) | 3 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Septic shock (Infections and infestations) | 2 | 2
Cellulitis (Infections and infestations) | 0 | 3
Gangrene (Infections and infestations) | 3 | 0
Influenza (Infections and infestations) | 1 | 2
Post procedural cellulitis (Infections and infestations) | 1 | 2
Infection (Infections and infestations) | 1 | 1
Post procedural infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Acute hepatitis B (Infections and infestations) | 1 | 0
American trypanosomiasis (Cardiac disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Ear infection (Cardiac disorders) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Graft infection (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Hepatobiliary infection (Infections and infestations) | 1 | 0
Infectious colitis (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Mediastinitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Post procedural pneumonia (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Puncture site infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 6
Gastritis (Gastrointestinal disorders) | 3 | 3
Colitis (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Diverticulum (Gastrointestinal disorders) | 2 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 3
Haematemesis (Gastrointestinal disorders) | 3 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 2
Duodenitis (Gastrointestinal disorders) | 1 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 2 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Proctitis ulcerative (Gastrointestinal disorders) | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Ulcerative gastritis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 19 | 15
Chest pain (General disorders) | 5 | 2
Death (General disorders) | 1 | 3
Multi-organ failure (General disorders) | 3 | 0
Chest discomfort (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Vascular stent restenosis (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Catheter site haematoma (General disorders) | 0 | 1
Catheter site haemorrhage (General disorders) | 1 | 0
Discomfort (General disorders) | 1 | 0
Drug intolerance (Gastrointestinal disorders) | 1 | 0
Medical device complication (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 | 7
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 3
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 2 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 3 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0
Postoperative renal failure (Injury, poisoning and procedural complications) | 0 | 2
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Failure to anastomose (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Graft loss (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hepatic rupture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Postimplantation syndrome (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 13
Chronic kidney disease (Renal and urinary disorders) | 3 | 6
Renal failure (Renal and urinary disorders) | 1 | 4
Haematuria (Renal and urinary disorders) | 2 | 2
Calculus ureteric (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Renal impairment (Renal and urinary disorders) | 1 | 1
Urogenital haemorrhage (Renal and urinary disorders) | 1 | 1
Bladder tamponade (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1
Renal haematoma (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Hypotension (Vascular disorders) | 5 | 4
Hypertension (Vascular disorders) | 4 | 2
Peripheral ischaemia (Vascular disorders) | 6 | 0
Haematoma (Vascular disorders) | 0 | 4
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 1
Hypertensive crisis (Vascular disorders) | 1 | 2
Circulatory collapse (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 1
Air embolism (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1
Arterial haemorrhage (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Artery dissection (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Ischaemia (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Troponin increased (Investigations) | 11 | 9
Laboratory test abnormal (Investigations) | 3 | 1
Troponin I increased (Investigations) | 2 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1
Troponin T increased (Investigations) | 2 | 1
Hepatic enzyme increased (Investigations) | 1 | 1
Liver function test abnormal (Investigations) | 1 | 1
Myocardial necrosis marker increased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Electrocardiogram change (Investigations) | 1 | 0
Haemoglobin abnormal (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 | 0
Back disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 5 | 4
Carotid artery stenosis (Nervous system disorders) | 4 | 0
Dizziness (Nervous system disorders) | 3 | 1
Paraesthesia (Nervous system disorders) | 2 | 1
Encephalopathy (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Brain stem haemorrhage (Nervous system disorders) | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Quadranopia (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Vertebral artery stenosis (Nervous system disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 2
Cholecystitis acute (Hepatobiliary disorders) | 4 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic ischaemia (Hepatobiliary disorders) | 1 | 0
Hepatic necrosis (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 1
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Blindness (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 3
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Primary hyperaldosteronism (Endocrine disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1752) | Losmapimod 7.5 mg BID (N=1724)
Hypertension (Vascular disorders) | 49 | 33
Hypotension (Vascular disorders) | 29 | 36
Troponin increased (Investigations) | 39 | 23
Angina pectoris (Cardiac disorders) | 32 | 40
Atrial fibrillation (Cardiac disorders) | 65 | 72
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 47
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 61 | 48
Anemia (Blood and lymphatic system disorders) | 35 | 39
Dizziness (Nervous system disorders) | 37 | 39
Non-cardiac chest pain (General disorders) | 41 | 44
Diarrhoea (Gastrointestinal disorders) | 41 | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.